CLINICAL TRIAL: NCT06828445
Title: Increasing Use of SNAP Fruit and Vegetable Incentive Programs for Families With Food Insecurity
Brief Title: Increasing Affordable Fruits and Vegetables for Families With Food Insecurity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Virginia Commonwealth University (Other); Cornell University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Adams, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00136502; R01DK140677 (NIH)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Diet
Keywords: food insecurity; diet; Supplemental Nutrition Assistance Program; fruit; vegetable; healthy eating; pediatrician

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet intervention (Experimental): Caregivers will receive brief education about a SNAP fruit and vegetable incentive program in South Carolina during their child's pediatrician visit. Following the visit, caregivers will receive a "free trial" of this SNAP program to encourage first-time use. After the free trial, caregivers can continue purchasing the same fruit and vegetable boxes at a steeply discounted price using their SNAP card. Free home delivery during the "free trial" and for all subsequent boxes purchased at a discounted rate will be offered during the full study duration.
  Interventions: Behavioral: Veggie Vouchers
- Education-only wait-list control (No Intervention): Caregivers will only receive brief education about a SNAP fruit and vegetable incentive program in South Carolina during their child's pediatrician visit. Once caregivers complete all study measures, they will be moved off the wait list and offered the intervention.

INTERVENTIONS:
Behavioral: Veggie Vouchers — Caregivers will receive brief education about a SNAP fruit and vegetable incentive program in South Carolina during their child's pediatrician visit. Following the visit, caregivers will receive a "free trial" of this SNAP program to encourage first-time use. After the free trial, caregivers can continue purchasing the same fruit and vegetable boxes at a steeply discounted price using their SNAP card. Free home delivery during the "free trial" and for all subsequent boxes purchased at a discounted rate will be offered during the full study duration.
  Arms: Diet intervention

SUMMARY:
Investigator will test an intervention to increase use of a fruit and vegetable incentive program in South Carolina for families in the Supplemental Nutrition Assistance Program (SNAP) experiencing food insecurity. Caregivers are randomized to an intervention or an education-only, wait-list control group. The investigators hypothesize the intervention will improve diet-related outcomes, above and beyond the education-only wait-list control.

DETAILED DESCRIPTION:
This study will test an intervention to increase use of a fruit and vegetable incentive program for families in the Supplemental Nutrition Assistance Program (SNAP) using a randomized controlled trial design. Caregivers are randomized to the intervention or an education-only wait-list control group. All caregivers are given brief education about a SNAP fruit and vegetable incentive program. Caregivers in the intervention are also given an initial "free trial" of this program and free home delivery. The primary aim is to examine intervention efficacy on diet-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver 18+ years of age
* Has a child 2-10 years of age
* Speaks English
* Screens positive for food insecurity
* Currently enrolled in the Supplemental Nutrition Assistance Program (SNAP)
* Lives with a feasible radius for home delivery
* Consistent access to a phone that receives text messages

Exclusion Criteria:

* Anticipate no longer being enrolled in SNAP during the study duration
* Recent use of the SNAP fruit and vegetable incentive program
* Caregiver or child has a medical condition that impacts their ability to eat fruits and vegetables
* Caregiver or child has a significant food allergy, preference, or intolerance that impacts their ability to eat fruits and vegetables

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 296 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Child diet quality | Baseline, 6, 18, and 30 weeks
  Caregivers will complete a 3-day food record for their child's dietary intake. Child diet quality will then be assessed using the Healthy Eating Index.

SECONDARY OUTCOMES:
Caregiver diet quality | Baseline, 6, 18, and 30 weeks
  Caregivers will complete a 3-day food record for their dietary intake. Caregiver diet quality will then be assessed using the Healthy Eating Index.
Child Eating Behaviors | Baseline, 6, 18, and 30 weeks
  The Children's Eating Behavior Questionnaire will be used to assess children's food fussiness. The food fussiness sub-scale consists of 5-pt Likert scale items ranging from Never (1) to Always (5). The mean of the response values is calculated. Higher score indicating a greater degree of food fussiness.
Process metrics | Through study completion, an average of 3 years
  Process metrics will examine the reach of families who received brief education during clinic visits at each site, utilization of the free trial, use of home delivery, and families who cycled off SNAP within the study duration (%, #, timing).
Intervention utilization | Through study completion, an average of 3 years
  Semi-structured phone interviews and surveys will be administered to caregivers to elicit perceptions on intervention components, barriers/facilitators to intervention use, and suggestions for future dissemination.
Perspectives of the intervention | Through study completion, an average of 3 years
  Focus groups and online surveys will be administered to key informants to assess barriers and facilitators to intervention implementation and sustainability.
Food security | Baseline, 6, 18, and 30 weeks
  The United States Department of Agriculture Household Food Security Module (18-item) will be administered. Higher scores indicate less food security.
Availability Pillar of Food Security | Baseline, 6, 18, and 30 weeks
  The Perceived Limited Availability scale will be administered (6-items). Items are summed to create a total score for food stores (3-items) and food pantries (3 items). Each total score ranges 0-3. Higher scores are considered less desirable.
Utilization Pillar of Food Security | Baseline, 6, 18, and 30 weeks
  The Utilization Barriers scale (8-items) will be administered. Items are summed to create a score ranging 0-8. Higher scores are considered less desirable.
Stability Pillar of Food Security | Baseline, 6, 18, and 30 weeks
  The Food Insecurity Stability scale (12-items) will be administered. Participants receive 4 scores, each ranging from 0-3 for chronic, seasonal, monthly, and intermittent food insecurity. Higher scores indicate a greater degree of chronic, seasonal, monthly, and intermittent food insecurity.
Nutrition Security | Baseline, 6, 18, and 30 weeks
  Nutrition security will be measured using the Household Nutrition Security scale (4-items). Item scores range 0 ("Always") to 4 ("Never"). The mean of item scores is calculated. Higher scores indicate a greater degree of nutrition security.
Household Healthfulness Choice | Baseline, 6, 18, and 30 weeks
  The Household Healthfulness Choice (3-items) survey will be administered. Items are scored from 4 ("Always") to 0 ("Never"). The mean of the item scores is calculated. Higher scores indicate a greater degree healthfulness choice.
Dietary Choice | Baseline, 6, 18, and 30 weeks
  The Dietary Choice (3-items) survey will be administered. Item scores range from 0 ("Always") to 4 ("Never"). The mean of the item scores is calculated. Higher scores indicate a greater degree of dietary choice.
SNAP fruit and vegetable incentive program utilization | Through study completion, an average of 3 years
  Purchasing data will be used to quantify the number and type of produce boxes purchased as part of the Supplemental Nutrition Assistance Program (SNAP) fruit and vegetable incentive program in South Carolina.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No